CLINICAL TRIAL: NCT05844332
Title: LUTATHERA Injection General Use Result Survey (Somatostatin Receptor-positive Neuroendocrine Tumor, CAAA601A11401)
Brief Title: LUTATHERA Injection General Use Result Survey
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA601A11401
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Somatostatin Receptor-positive Neuroendocrine Tumor
Keywords: LUTATHERA
MeSH Terms: interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- LUTATHERA: patients treated with LUTATHERA Injection
  Interventions: Other: LUTATHERA

INTERVENTIONS:
Other: LUTATHERA — There was no treatment allocation. Patients administered LUTATHERA by prescription could be enrolled.
  Other Names: Lutetium oxodotreotide (177Lu)

SUMMARY:
This study was a multicenter observational study with a central registration system and all-case surveillance system without a control group.

DETAILED DESCRIPTION:
From the date of the first dose of this drug until 40 weeks after the date of the last dose (64 weeks if 4 doses are administered 8 weeks apart).

For patients who discontinue treatment with this drug during the observation period, necessary variables were examined until 40 weeks after the last dose of this drug during the observation period and recorded in the case report forms (CRF).

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with this drug for the following indications during a certain post-marketing period

  * Indication: Somatostatin receptor-positive neuroendocrine tumor Patients who started to receive this drug before the contract for this study will also be included in the study population and it will be allowed to register them after the contract so that all patients who receive this drug will be included in this study. Patients treated with this drug for off-label indication will also be included in this study to register all patients received this drug.

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with this drug for the following indications during a certain post-marketing period
  • Indication: Somatostatin receptor-positive neuroendocrine tumor
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Renal dysfunction, Myelosuppression, Myelodysplastic syndrome/acute myeloid leukaemia and Hormone release induced crises | Until 40 weeks after the date of the last dose (64 weeks if 4 doses are administered 8 weeks apart).
  To evaluate the safety about Renal dysfunction, Myelosuppression, Myelodysplastic syndrome/acute myeloid leukaemia and Hormone release induced crises after administration of this drug in a real world setting

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- Japan (43):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Hirosaki, Aomori
  - Novartis Investigative Site, Kamogawa, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukui-shi, Fukui
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Iwata, Shizuoka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18390